CLINICAL TRIAL: NCT04116177
Title: Flexible vs. Standard Programming in Parkinson's Disease Patients Receiving Subthalamic Implant: a Double-blind Cross-over Trial
Brief Title: Flexible vs. Standard Deep Brain Stimulation Programming in Parkinson Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Alfonso Fasano, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 15-9700
Record Dates: First submitted 2019-09-25; First posted 2019-10-04 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Parkinson Disease
Keywords: Deep brain stimulation; Parkinson disease; Novel strategies
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Stimulation (Active Comparator): Standard stimulation using contact 3-6 to achieve best therapeutic stimulation
  Interventions: Device: Deep brain stimulation
- Flexible stimulation (Experimental): Flexible stimulation using all available stimulation strategies provided by the VerciseTM system including stimulation of contacts 1-8 and variable pulse width and frequency.
  Interventions: Device: Deep brain stimulation

INTERVENTIONS:
Device: Deep brain stimulation — Stimulation using VerciseTM system

SUMMARY:
Exploring the benefits of the linear lead in deep brain stimulation.

DETAILED DESCRIPTION:
Detailed Description:

This is a single-centre, double-blinded cross-over study comparing the 4 contact vs 8 contact electrodes of deep brain stimulation (DBS) patients.

The study will follow 2 phases.

Phase 1:

Visit 1 Screening/Baseline (T0):

As per current standard care for patients undergoing subthalamic deep brain stimulation (STN-DBS), participants will be screened 3-6 months before the surgery (T0) according to the inclusion/exclusion criteria.

Visits for standard programming of VerciseTM system between 1 to 3 months after the surgery of 10 patients will be done in an open label fashion in order to find the best program for optimization of patient motor symptoms without side effects. This will be done according to the standard of practice currently adopted at Toronto Western Hospital.

Phase 2:

Visit 1

Randomization: 4 months +/- 4weeks of the surgery, patients will be randomized to two type of stimulation:

1. Standard : only contacts 3-6 will be used in either unipolar or bipolar configuration; pulse width lower than 60μsec will not be used; all types of frequencies will be used but keeping the value constant for the both hemispheres at each active contact. The same amount of current for each of the active contacts will be used, however, in case of different currents at different contacts, an "interleaved" type of stimulation will be used and frequency will kept lower than 125Hz ( Fig 2A).
2. Flexible : contacts 1-8 will be used in any possible configuration and using different amount of current for each of the active one as well as different frequencies; pulse width lower than 60μsec can be used. In conclusion, all the capabilities of the VerciseTM system will be used. Possible adjustments to stimulation parameters (e.g. Pulse width, amplitude threshold) will be performed to achieve an optimal therapeutic window for each patient.

Visit 2

Follow up visit at 6 months +/- 4 weeks of the surgery for neurological examination if required.

Visit 3 (T1):

Cross over : 7 months +/- 4 weeks after the surgery patients will be switched to the other type of stimulation . Raters and patients will be blinded to the group allocation.

Visit 4:

Follow up visit at 9 months +/- 4 weeks of the surgery for neurological examination if required.

Visit 5 (T2):

End of study visit at month 10 +/- 4 weeks after the surgery. Raters and patients will be blinded to the group allocation.

There might be unscheduled visits in case of unexpected clinical conditions (i.e. occurrence of side effects or worsening of motor conditions). Participants will be in this study for a maximum of 17 months. Throughout the whole study, participants will visit the clinic without their regular medication for PD as part of standard treatment practice. All the stimulation adjustment will be performed by the same unblinded physician using the GuideTM software provided by the company.

ELIGIBILITY:
Inclusion Criteria:

1) Patients with a diagnosis of PD according to the British Parkinson's Disease Society

1. Brain Bank criteria (Hughes, Daniel, Kilford, & Lees, 1992), who fulfilled the inclusion and exclusion criteria proposed by the core assessment programme for surgical interventional therapies in PD panel (Defer, Widner, Marié, Rémy, & Levivier, 1999)
2. Male and female patients with idiopathic PD, who have symptoms responsive to L-dopa medications, but who have significant impairment related to PD that is no longer well controlled with pharmacotherapy (i.e., refractory to optimized medical therapy)
3. Patients considered as STN-DBS candidates as per current standard of care. These patients will subsequently undergo STN-DBS surgery and maintain stimulation therapy.
4. Quality of life and social functioning influenced by levodopa-responsive signs
5. No major comorbidities

Exclusion Criteria:

1) Exclusion criteria will include patients with other significant neurologic or psychiatric illnesses or cognitive deficit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Change of Overall Global functioning (PGIC) | After 3 months of each intervention
  The PGIC evaluates all aspects of patients' health and assesses if there has been an improvement or decline in clinical status relative to baseline. This is a seven point scale with lower values indicating worsening and higher values, improvement.

SECONDARY OUTCOMES:
Measure of Quality of life (PDQ-39) | After 3 months of each intervention
  The PDQ-39 assesses individuals experiences across 8 dimensions of daily living. Each dimension is scored from 0 to 100. Lower scores mean better quality of life.
Clinical change in motor symptoms using Unified Parkinson Disease Rating Scale I-IV | After 3 months of each intervention
  The Unified Parkinson Disease Rating Scale I-IV ranges from 0-199, with higher scores meaning more severe disease
Clinical change in motor symptoms | After 3 months of each intervention
  Clinical change in motor symptoms as measured using falls diaries
Number of falls | After 3 months of each intervention
  Using a falls diary
Change in the presence and severity of depressive symptoms using the Beck Depression Inventory (BDI) | After 3 months of each intervention
  The BDI is a 21-question multiple-choice self-report inventory for measuring the severity of depression. Scores range from 0 to 63, with higher scores meaning worse depression.
Walking speed measure using Prokinetics gait analysis/Zeno Walkway | After 3 months of each intervention
  The Zeno Walkway is a 20 feet walking mat containing 16-pressure sensing pads and circuitry that allows for measurement of various gait and balance variables during straight walking. Patients will be asked to walk on the mat at a self selected pace. Walking speed will be measured.
Step length measured using Prokinetics gait analysis/Zeno Walkway | After 3 months of each intervention
  The Zeno Walkway is a 20 feet walking mat containing 16-pressure sensing pads and circuitry that allows for measurement of various gait and balance variables during straight walking. Patients will be asked to walk on the mat at a self selected pace. Mean and coefficients of variation (standard deviation divided by the mean x 100) of step length will be measured.
Cadence measured using Prokinetics gait analysis/Zeno Walkway | After 3 months of each intervention
  The Zeno Walkway is a 20 feet walking mat containing 16-pressure sensing pads and circuitry that allows for measurement of various gait and balance variables during straight walking. Patients will be asked to walk on the mat at a self selected pace. Mean and coefficients of variation (standard deviation divided by the mean x 100) of cadence will be measured. Cadence is the number of steps per minute of walking.
Double support time measured using Prokinetics gait analysis/Zeno Walkway | After 3 months of each intervention
  The Zeno Walkway is a 20 feet walking mat containing 16-pressure sensing pads and circuitry that allows for measurement of various gait and balance variables during straight walking. Patients will be asked to walk on the mat at a self selected pace. Mean and coefficients of variation (standard deviation divided by the mean x 100) of double support time will be measured. The double support time is the the time during gait where both feet are in contact to the ground

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Movement disorders Centre, Toronto Western Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fasano A, Daniele A, Albanese A. Treatment of motor and non-motor features of Parkinson's disease with deep brain stimulation. Lancet Neurol. 2012 May;11(5):429-42. doi: 10.1016/S1474-4422(12)70049-2. PMID 22516078
- [Background] Herzog J, Pinsker M, Wasner M, Steigerwald F, Wailke S, Deuschl G, Volkmann J. Stimulation of subthalamic fibre tracts reduces dyskinesias in STN-DBS. Mov Disord. 2007 Apr 15;22(5):679-84. doi: 10.1002/mds.21387. PMID 17266046
- [Background] Herzog J, Hamel W, Wenzelburger R, Potter M, Pinsker MO, Bartussek J, Morsnowski A, Steigerwald F, Deuschl G, Volkmann J. Kinematic analysis of thalamic versus subthalamic neurostimulation in postural and intention tremor. Brain. 2007 Jun;130(Pt 6):1608-25. doi: 10.1093/brain/awm077. Epub 2007 Apr 17. PMID 17439979
- [Background] Chastan N, Westby GW, Yelnik J, Bardinet E, Do MC, Agid Y, Welter ML. Effects of nigral stimulation on locomotion and postural stability in patients with Parkinson's disease. Brain. 2009 Jan;132(Pt 1):172-84. doi: 10.1093/brain/awn294. Epub 2008 Nov 11. PMID 19001482
- [Background] Weiss D, Walach M, Meisner C, Fritz M, Scholten M, Breit S, Plewnia C, Bender B, Gharabaghi A, Wachter T, Kruger R. Nigral stimulation for resistant axial motor impairment in Parkinson's disease? A randomized controlled trial. Brain. 2013 Jul;136(Pt 7):2098-108. doi: 10.1093/brain/awt122. Epub 2013 Jun 11. PMID 23757762
- [Background] Barbe MT, Maarouf M, Alesch F, Timmermann L. Multiple source current steering--a novel deep brain stimulation concept for customized programming in a Parkinson's disease patient. Parkinsonism Relat Disord. 2014 Apr;20(4):471-3. doi: 10.1016/j.parkreldis.2013.07.021. Epub 2013 Sep 14. No abstract available. PMID 24041939
- [Background] Hoehn MM, Yahr MD. Parkinsonism: onset, progression and mortality. Neurology. 1967 May;17(5):427-42. doi: 10.1212/wnl.17.5.427. No abstract available. PMID 6067254
- [Background] Jenkinson C, Fitzpatrick R, Peto V, Greenhall R, Hyman N. The Parkinson's Disease Questionnaire (PDQ-39): development and validation of a Parkinson's disease summary index score. Age Ageing. 1997 Sep;26(5):353-7. doi: 10.1093/ageing/26.5.353. PMID 9351479
- [Background] Timmermann L, Jain R, Chen L, Maarouf M, Barbe MT, Allert N, Brucke T, Kaiser I, Beirer S, Sejio F, Suarez E, Lozano B, Haegelen C, Verin M, Porta M, Servello D, Gill S, Whone A, Van Dyck N, Alesch F. Multiple-source current steering in subthalamic nucleus deep brain stimulation for Parkinson's disease (the VANTAGE study): a non-randomised, prospective, multicentre, open-label study. Lancet Neurol. 2015 Jul;14(7):693-701. doi: 10.1016/S1474-4422(15)00087-3. Epub 2015 May 28. PMID 26027940